CLINICAL TRIAL: NCT01444248
Title: A Multi-center, Open, Randomized, Parallel-group Study to Compare the Compliance of Patients Treated With Once-daily (od) or Twice-daily (Bid) Glimepiride and Metformin Fixed Combination Therapy
Brief Title: Compare the Compliance of Patients Treated With Once-daily (od) or Twice-daily (Bid) Glimepiride and Metformin Fixed Combination Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HANDOK2009.02
Record Dates: First submitted 2011-09-21; First posted 2011-09-30 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Amaryl MEX
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amaryl MEX (Experimental)
  Interventions: Drug: Glimepiride/ Metformin
- Amaryl M (Active Comparator)
  Interventions: Drug: Glimepiride/ Metformin

INTERVENTIONS:
Drug: Glimepiride/ Metformin — 4/1000mg once daily
  Arms: Amaryl MEX
Drug: Glimepiride/ Metformin — 4/1000mg bid
  Arms: Amaryl M

SUMMARY:
The study design of this trial is open-label, randomized, multi-center, parallel-group study.

DETAILED DESCRIPTION:
The effectiveness of treatment of a disease depends mainly on two factors: the efficacy of the treatment and the compliance of the patient with this treatment. Polymedication is one of the predisposing factors to low compliance in type 2 DM. It can be expected that a simple regimen may improve compliance. Amaryl Mex phase III trial was not designed to compare the compliance of patients with different dosing regimens of oral antidiabetic drugs. However, it was found that patients' compliance in the morning was better than in the evening, suggesting that Amaryl Mex once daily regimen may improve compliance. Pill count is the gold standard for measuring compliance, but this method provides incomplete and unreliable results. Advanced electronic monitoring device obtains details of patients' behavior during the day and over long periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 ~ 75 years at screening
* Patients who have been diagnosed with type 2 DM for at least 3 months
* Patients who were treated with a stable dose with combination therapy of glimepiride 4mg or more and metformin 1000mg or more which can switch to Amaryl M 2/500mg bid or Amaryl Mex 2/500mg 2T od regimen.
* HbA1c ≤ 9 % at randomization
* BMI ≤ 40 kg/m2 at randomization
* Patients who would give the informed consent
* Patients who can perform SMBG and record the data on the patient's diary
* Patients who can understand and use MEMS properly

Exclusion Criteria:

* Patients with the medical history of acute metabolic complications such as diabetic ketoacidosis, hyperosmolar nonketotic coma within 3 months prior to the study participation
* Patients who are under insulin therapy at randomization
* Patients who received systemic corticosteroid agent within 4 weeks prior to the study participation
* Patients with acute, severe cardiovascular disease (e.g., heart failure, myocardial infarction, stroke, etc).
* Pregnant or lactating females
* history of drug or alcohol abuse
* Patients with known hypersensitivity to the ingredient of the study drug or drugs in sulfonylurea, sulfonamide, biguanide class
* Night-shift workers
* Patients with an experience of participating in other clinical trial within 3 months prior to the study participation
* Clinically significant laboratory abnormality on screening labs or any medical condition that would affect the completion or outcome of the study based on investigator's decision
* Patients with serum creatinine level > 1.5 mg/dl in male and > 1.4 mg/dl in female
* Patients with ALT or AST > 3x ULN
* Any conditions requiring help of others with drug administration (e.g. manual disability, serious visual defect, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
compliance of patients treated with once-daily or twice-daily | 24 weeks

SECONDARY OUTCOMES:
Blood glucose lowering effect | 24 weeks
Episodes of hypoglycaemia | 24 weeks
other adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sungwoo Park, professor, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Handok Pharmaceuticals, Seoul, Seoul, South Korea